CLINICAL TRIAL: NCT05440396
Title: Development of an Artificial Intelligence Model of Image Recognition Through Images of Intravascular Catheters From Inpatients and Outpatients to Identify the Presence of Local Signs Associated With Infection
Brief Title: Identifying Local Signs at the Catheter Insertion Site With Artificial Intelligence
Acronym: DeepCath
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Outcome Rea (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other); National Network Surveillance and Prevention of Infections Associated with Invasive Devices SPIADI (Unknown); University Hospital, Clermont-Ferrand (Other); University Hospital, Grenoble (Other); UNICANCER (Other); University Grenoble Alps (Other)
Responsible Party: Sponsor
Other Study IDs: DeepCath
Record Dates: First submitted 2022-06-21; First posted 2022-06-30 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Catheter Infection
Keywords: catheter infection; deep learning; local signs
MeSH Terms: interventions — Growth and Development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patient: Patients will be recruited independently in each of the centers participating in the study, according to the specific organization of each service (hospital and home). Patients will be selected based on the study inclusion/non-inclusion criteria. The included patients will receive oral information about the study. The informed consent will be obtained before any investigation.
  Each photograph will focus on the intravascular catheter. The investigators will respect the main non-inclusion criterion: not to show any peripheral identification sign close to the insertion point of the catheter that cannot be masked when the photograph is taken. In this context, jewellery, clothing, tattoos, scars, and birthmarks represent identifying features. Individual access accounts with secure, randomly generated passwords will be provided to investigators.
  The photographs will be anonymous, and any identification of the person concerned will be impossible.
  Interventions: Diagnostic Test: Photographs collection phase

INTERVENTIONS:
Diagnostic Test: Photographs collection phase — Three medical experts have been selected to review the photo collected. Each expert medical assesses the presence of local signs of infection on the photographs by annotating them directly via a dedicated software. They will annotate local signs: redness, perfusion extravasation, necrosis, hematoma, edema, non-purulent discharge, and purulent discharge.
  A convolutional neural network model will determine the probability of local sign presence. Each picture will be annotated to determine the main characteristics of the catheter. A dataset preparation with photo cropping will be performed for modelling.
  Other Names: Photographs reviewing phase by medical experts; Development/Validation of artificial intelligence algorithm

SUMMARY:
Deepcath is the first step to the introduction of artificial intelligence in catheter care. A better use of visualisation of catheter exit site should be used not only by the HCWs but also by the patients and their family.

A deep learning system able to detect visual abnormalities of the catheter exit site will be an helpful tools to develop a continuous follow-up of intravascular catheters.

ELIGIBILITY:
Inclusion Criteria:

Patients over 18 years of age Patients with one or more implanted central venous, midline, piCCline, arterial, or peripheral catheters.

Patient and/or trusted person and/or family who have verbally stated their non-objection to the study Patient affiliated or beneficiary of a social security plan

Exclusion Criteria:

Patients presenting a peripheral identification sign close to the catheter insertion point cannot be masked when the photograph is taken. Thus, jewelry, clothing, tattoos, scars, and birthmarks are identifying features.

Patients whose catheter insertion point is not visible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited independently in each of the centers participating in the study, according to the specific organization of each service (hospital and home). Patients will be selected based on the study inclusion/non-inclusion criteria. The included patients will receive oral information about the study. The informed consent will be obtained before any investigation.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of correct predictions for redness divided by the total number of predictions | through study completion, an average of 1 year
  Overall classification accuracy of the learning model compared to the assessment of three independent medical experts on the detection of the presence of redness greater than or equal to 5 mm at the catheter insertion site.

SECONDARY OUTCOMES:
The ratio of true positives and total positives predicted: | through study completion, an average of 1 year
  The precision metric focuses on Type-I errors(FP). A Type-I error occurs when we reject a true null Hypothesis.
The number of correct predictions for indurated venous cord divided by the total number of predictions | through study completion, an average of 1 year
  Evaluate, on the basis of images of peripheral catheter insertion sites, the reliability of the learning model on the assessment of the presence of indurated venous cord.
The link between presence of local signs and infection | through study completion, an average of 1 year
  Measure the correlation between the appearance of the catheter puncture site and the presence of signs consistent with local and systemic infection.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François TIMISIT, Pr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (4):
- France (4):
  - CHU Grenoble Alpes, Grenoble, Isère
  - CHU Clermont-Ferrand, Clermont-Ferrand, Puy-de-Dôme
  - Réseau RéPIAS SPIADI, Tours
  - Hôpital Bichat - Claude-Bernard, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Timsit JF, Schwebel C, Bouadma L, Geffroy A, Garrouste-Orgeas M, Pease S, Herault MC, Haouache H, Calvino-Gunther S, Gestin B, Armand-Lefevre L, Leflon V, Chaplain C, Benali A, Francais A, Adrie C, Zahar JR, Thuong M, Arrault X, Croize J, Lucet JC; Dressing Study Group. Chlorhexidine-impregnated sponges and less frequent dressing changes for prevention of catheter-related infections in critically ill adults: a randomized controlled trial. JAMA. 2009 Mar 25;301(12):1231-41. doi: 10.1001/jama.2009.376. PMID 19318651
- [Result] Timsit JF. Diagnosis and prevention of catheter-related infections. Curr Opin Crit Care. 2007 Oct;13(5):563-71. doi: 10.1097/MCC.0b013e3282efa03f. PMID 17762237
- [Result] Buetti N, Rickard CM, Timsit JF. Catheter dressings. Intensive Care Med. 2022 Aug;48(8):1066-1068. doi: 10.1007/s00134-022-06734-w. Epub 2022 May 27. No abstract available. PMID 35624170
- [Result] Blot S, Ruppe E, Harbarth S, Asehnoune K, Poulakou G, Luyt CE, Rello J, Klompas M, Depuydt P, Eckmann C, Martin-Loeches I, Povoa P, Bouadma L, Timsit JF, Zahar JR. Healthcare-associated infections in adult intensive care unit patients: Changes in epidemiology, diagnosis, prevention and contributions of new technologies. Intensive Crit Care Nurs. 2022 Jun;70:103227. doi: 10.1016/j.iccn.2022.103227. Epub 2022 Mar 3. PMID 35249794
- [Result] Buetti N, Mermel LA, Timsit JF. Routine catheter-tip cultures for assessing catheter-related bloodstream infections in randomised-controlled trials. Anaesth Crit Care Pain Med. 2022 Feb;41(1):101006. doi: 10.1016/j.accpm.2021.101006. Epub 2021 Dec 14. No abstract available. PMID 34920150
- [Result] Buetti N, Abbas M, Pittet D, Chraiti MN, Sauvan V, De Kraker MEA, Boisson M, Teixeira D, Zingg W, Harbarth S. Lower risk of peripheral venous catheter-related bloodstream infection by hand insertion. Antimicrob Resist Infect Control. 2022 Jun 3;11(1):80. doi: 10.1186/s13756-022-01117-8. PMID 35659775